CLINICAL TRIAL: NCT01405248
Title: Butylphthalide for Preventing Restenosis After Intracranial and Extracranial Artery Stenting
Acronym: BPRIAS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jinling Hospital, China (Other)
Collaborators: CSPC-NBP Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Xinfeng Liu, Butylphthalide for Preventing Restenosis After Intracranial and Extracranial Artery Stenting, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BPRIAS
Record Dates: First submitted 2011-07-28; First posted 2011-07-29 (Estimated); Last update posted 2015-10-26 (Estimated); Status verified 2015-10

CONDITIONS: Restenosis
Keywords: Butylphthalide
MeSH Terms: interventions — 3-n-butylphthalide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Butylphthalide (Experimental): Single center of the placebo control a double-blind randomized control study to evaluate Butylphthalide prevention stents restenosis effect
  Interventions: Drug: Butylphthalide
- control (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Butylphthalide — 20 mg/time per os three times a day. 180days
  Other Names: NBP
  Arms: Butylphthalide
Drug: Placebo — 20 mg/time per os three times a day. 180days
  Arms: control

SUMMARY:
The purpose of this study is to determine whether butylphthalide are effective for Preventing Restenosis after Intracranial and Extracranial Artery Stenting

DETAILED DESCRIPTION:
Ischemic stroke is a significant cause of death, most of the patients is caused by atherosclerosis,current treatments include internal medicine medications, interventional treatment and so on,among them, the interventional therapy can make narrow blood vessels blood recovery fastly,and for its small trauma,Gradually accepted by psychiatrist, But stents are easy to narrow has been plagued by everybody ,At present, prevent restenosis stent is mainly of antiplatelet therapy,But,prevention effect is not obvious often easy to appear harmful response,how to effectively reduce postoperative restenosis, become the majority concern of patients and doctors .Clinical trials showed that, butylbenzene can promote the function of ischemic stroke recovery patients. Animal pharmacodynamics study suggests that this product can block the ischemic stroke of brain damage caused by DuoGe pathological link, with strong against ischemic and brain protection, especially can obviously increase in small brains ischemia ATP and phosphoric acid creatine level, decrease local cerebral ischemia in rats, reduce infarct size, cerebral edema improved energy metabolism and brain ischemia of microcirculation and blood flow in the brain, restrain the nerve cell apoptosis, and has the cerebral thrombosis and anti-platelet aggregation function. Research shows that, butylbenzene phthalocyanine influence through arachidonic acid (AA) metabolism, selective inhibition and their metabolites from DuoZhong mediated pathophysiological events, can remove microvascular spasms. Inhibit platelet aggregation, restrain TXA2 synthesis, scavenging free radicals, thereby through many ways, many link blocking caused by cerebral ischemia the pathophysiology of development process. These mechanisms may make butylbenzene in preventing phthalocyanine intracranial carotid stenting noted restenosis and related ischemia of events play an important role.

ELIGIBILITY:
Inclusion Criteria:

1. . DSA check to be sure, the VA, BA ICA, MCA, PCA and other major blood vessels, have corresponding stenosis of symptoms more than 50%, not corresponding symptoms stenosis of greater than 70%;
2. . A successful cerebrovascular carotid stenting noted.

Exclusion Criteria:

1. . There is a serious bleeding tendency, nearly three months have intracranial bleeding or cranial out blood;
2. . Active peptic ulcer;
3. . Not good control high blood pressure; the wickedness of
4. . Blood vessel distortion, variation, narrow degree badly, can not be implemented stents operation;
5. . Serious cardiopulmonary etc medical problems;
6. . Those allergic to celery;
7. . Contrast agents allergy;
8. . Can't complete follow-up.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-07; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
occlusion and restenosis | one year
  Stenosis detected by DSA(digital subtraction angiography), CTA(CT angiography) or MRA(MR angiography) was measured according to NASCET (North American Symptomatic Carotid Endarterectomy Trial) method.Concretely, NASCET stenosis is calculated from the ratio of the linear luminal diameter of the narrowest segment of the diseased portion of the artery to the diameter of the artery beyond any poststenotic dilatation: NASCET = (1-md/C)×100%.

SECONDARY OUTCOMES:
NIHSS, mRS | at one year
  NIHSS and mRS are widely used stroke deficit assessment tools. Most clinical stroke-related trials require a baseline and outcome severity assessment. The baseline of mRS is rank 0, NIHSS 0; the severity of mRS is 6, NIHSS 42. AS many patients have one or more strokes before they perform stening, this study selected NIHSS and mRS as the supplementary materials to estimate the stroke deficit of patients and to reflect the therapeutic effect and safety of stening and butylphthalide therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Xinfeng Liu, MD, Study Chair — Department of Neurology, Jinling Hospital, Nanjing University School of Medicine
Locations (1):
- Department of Neurology ;Jinling Hospital, Nanjing, Jiangsu, China